CLINICAL TRIAL: NCT04321395
Title: The Effect of Vigabatrin on Insulin Sensitivity
Brief Title: Vigabatrin and Insulin Sensitivity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202006177
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: NAFLD; Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity | interventions — Vigabatrin

STUDY DESIGN:
Intervention Model Description: Participants will receive vigabatrin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vigabatrin (Experimental)
  Interventions: Drug: Vigabatrin

INTERVENTIONS:
Drug: Vigabatrin — Vigabatrin - Pill, 500 mg twice daily for 7 days (days 0-6), 1000 mg twice daily for 7 days (days 7-13), 1500 mg twice daily for 10 days (days 14-23), 1000 mg twice daily for 7 days (days 24-30), 500 mg twice daily for 7 days (days 31-37) and will discontinue treatment on day 38.
  Other Names: sabril

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is a common complication of obesity and is associated with an increased risk of developing type 2 diabetes. The hallmark feature of NAFLD is an increase in intrahepatic triglyceride (IHTG) content. Data from studies conducted in rodent models suggest increased IHTG content can alter hepatic vagal afferent nerve (HVAN) activity. In rodent models of obesity and NAFLD, HVAN activity is reduced leading to impaired insulin sensitivity and glucose control. The reduction in HVAN activity is likely due to increased hepatic release of GABA, an inhibitory neurotransmitter, attributable to increased expression of GABA-Transaminase (GABA-T). Pharmacological inhibition of GABA-T in obese mice by treatment with vigabatrin, an irreversible inhibitor of GABA-T improves glucose tolerance and reduces hyperinsulinemia, hyperglycemia, and insulin resistance. It is not known if vigabatrin can also improve metabolic function in people. We propose to conduct a 3-week, single-arm trial to assess the effect size of treatment with vigabatrin on the following specific aims with the larger goal of determining whether a large, randomized controlled trial investigating the effect of vigabatrin is warranted.

ELIGIBILITY:
Inclusion Criteria:

* age 25-60 years old
* BMI 30.0-49.9 kg/m2
* IHTG content ≥5.6
* Homeostatic Model of Insulin Resistance (HOMA-IR) Score>2.5.

Exclusion Criteria:

* previous bariatric surgery
* structured exercise ≥250 min per week (e.g., brisk walking)
* unstable weight (>4% change during the last 2 months before entering the study)
* significant organ system dysfunction (e.g., diabetes, severe pulmonary, kidney or cardiovascular disease)
* cancer
* polycystic ovary syndrome
* major psychiatric illness (including suicidal ideation or previous suicide attempts)
* conditions that render subject unable to complete all testing procedures (e.g., severe ambulatory impairments, limb amputations, or metal implants that interfere with imaging procedures; coagulation disorders)
* regular use of tobacco products
* excessive consumption of alcohol (≥3 drinks/day for men and ≥2 drinks/day for women)
* use of medications that are known to affect the study outcome measures or increase the risk of study procedures and that cannot be temporarily discontinued for this study
* pre-existing visual field deficits; or those at high risk of irreversible vision loss, including patients with retinopathy or glaucoma
* pregnant or lactating women
* conditions that render subject unable to complete all testing procedures (e.g. aversion to needles, metal implants that prevent magnetic resonance imaging
* persons who are unable or unwilling to follow the study protocol
* persons who are not able to grant voluntary informed consent
* patients at risk for severe anemia (hemoglobin < 14 g/dL (men) or <12.0 g/dL (women) and/or hematocrit <40% in men or < 37% in women)
* patients with history of lower limb edema (risk of heart failure)
* patients with mild or more severe renal insufficiency (CrCl <100 mL/min (men) or <80 mL/min (women))
* patients with existing peripheral neuropathy
* women who have active menstrual cycles but are not using birth control (acceptable contraception includes barrier/hormonal/IUD)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vigabatrin
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vigabatrin
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4
Glucose infusion rate [Mean (Standard Deviation); unit: (mg/kg FFM/min)] | 6.61 (1.7)
2 Hour OGTT [Mean (Standard Deviation); unit: mg/dL] | 139.5 (7.9)
Oral Glucose Insulin Sensitivity [Mean (Standard Deviation); unit: ml/min/m^2 of body surface area] — Insulin sensitivity based on oral glucose tolerance. Values are calculated using glucose and insulin from a 3-hour 75 gram oral glucose tolerance test at 0, 2, and 3 hours. Higher values are indicate better insulin sensitivity.
  ml/min/m^2 of body surface area | 294 (56)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: Measured by hyperglycemic euglycemic clamp
Time Frame: 3 weeks after initiation of treatment
Measure: Mean (Standard Deviation); unit: mg/kg FFM/min
Arm/Group | Vigabatrin
Number analyzed (Participants) | 4
mg/kg FFM/min | 6.82 (1.7)

2. Secondary Outcome: Oral Glucose Tolerance
Description: Measured by 75 gram oral glucose tolerance test
Time Frame: 3 weeks after initiation of treatment
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Vigabatrin
Number analyzed (Participants) | 4
mg/dL | 155.5 (19.2)

3. Secondary Outcome: Oral Glucose Insulin Sensitivity
Description: Insulin sensitivity based on oral glucose tolerance. Values are calculated using glucose and insulin from a 3-hour 75 gram oral glucose tolerance test at 0, 2, and 3 hours. Higher values are indicate better insulin sensitivity.
Time Frame: After 3 weeks on drug
Measure: Mean (Standard Deviation); unit: ml/min/m^2 of body surface area
Arm/Group | Vigabatrin
Number analyzed (Participants) | 4
ml/min/m^2 of body surface area | 294 (56)

ADVERSE EVENTS:
Time Frame: Data were analyzed over the course of 6 months.
Description: Adverse events were assessed at each dose level.
Groups:
- Experimental: Vigabatrin: Vigabatrin: Vigabatrin - Pill, 500 mg twice daily for 7 days (days 0-6), 1000 mg twice daily for 7 days (days 7-13), 1500 mg twice daily for 10 days (days 14-23), 1000 mg twice daily for 7 days (days 24-30), 500 mg twice daily for 7 days (days 31-37) and will discontinue treatment on day 38.
Arm/Group | Experimental: Vigabatrin
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT04321395/Prot_SAP_000.pdf